CLINICAL TRIAL: NCT05006547
Title: Peroneal Muscles Response to Expected and Unexpected Falls Among Young and Middle-aged Adults Before and After Neuromuscular Training: a Cross Sectional-controlled Trial
Brief Title: Peroneal Muscles Response to Expected and Unexpected Falls Among Young and Middle-aged Adults Before and After Neuromuscular Training
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ariel University (Other)
Responsible Party: Sponsor
Other Study IDs: AU-HEA-SS-20210304:
Record Dates: First submitted 2021-07-21; First posted 2021-08-16 (Actual); Last update posted 2021-08-16 (Actual); Status verified 2021-03

CONDITIONS: Healthy Participants

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Young adults: 18<age<35
  Interventions: Other: Electromyograph Biofeedback training of the peroneal muscle
- Middle aged adults: 50<age<65
  Interventions: Other: Electromyograph Biofeedback training of the peroneal muscle

INTERVENTIONS:
Other: Electromyograph Biofeedback training of the peroneal muscle — The exercise will be performed with the subject sitting in front of a computer monitor, on an elevated chair, and his feet will be in the air. The examiner will ask the subject to perform a maximum contraction of the paronal muscles, in an open kinematic chain. After reference, the subject will begin a five-minute practice. The practice will be divided into rounds of: eight seconds of muscle work and 15 seconds rest.

SUMMARY:
Proper functioning of the ankle musculature, specifically peroneal muscles, is crucial for maintaining balance and reducing the risk for falls. Evidence suggests that a decrease in aspects of neuromuscular control already starts at midlife (45-65 years). However, there is almost no information regarding the function of the ankle muscles at the middle-age as most experiments have compared young (<35 years) and older subjects (>65 years). Moreover, neuromuscular training can improve the function of ankle muscle in response to perturbation; yet, no previous study has compared the level of effectiveness between middle-aged and young adults.

ELIGIBILITY:
Inclusion Criteria:

- Healthy participants

Exclusion Criteria:

* Neurological disease accompanied by motor, sensory or cognitive impairment.
* Illness or condition that does not allow strenuous activity.
* Significant orthopedic injury to the back or lower limbs in the last six months, which limits strenuous activity or weight-bearing.
* History of orthopedic injury that includes injury to the knee or ankle ligaments.
* Taking medications that may affect stability or balance. Significant visual impairment that is not corrected using glasses/contact lenses
* Pregnancy

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy participants- Twenty-five middle-aged (50-65years) and 25 young adults (20-35 years) will be recruited.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2021-07-01 (Actual); Primary Completion 2022-07-01 (Estimated); Study Completion 2022-07-01 (Estimated)

PRIMARY OUTCOMES:
Time to stabilization | Within 24 hours
  Subjects will be asked to jump from a 20 cm high box onto a force plate (i.e., expected fall).
Electromyography of peroneus longus- "The height of the amplitude"- expected fall | Within 24 hours
  Subjects will be asked to jump from a 20 cm high box onto a force plate (i.e., expected fall). electromyography of peroneus longus will be measured the height of the amplitude - expresses the peak of the electrical activity of the muscles.
Electromyography of peroneus longus- "Time to Peak"- expected fall | Within 24 hours
  Subjects will be asked to jump from a 20 cm high box onto a force plate (i.e., expected fall). electromyography of peroneus longus will be measured the "Time to Peak"- describes the time it takes for the Peroneus longus muscle to reach the peak of its electrical activity.
Electromyography of peroneus longus- "Time to Onset"- expected fall | Within 24 hours
  Subjects will be asked to jump from a 20 cm high box onto a force plate (i.e., expected fall). electromyography of peroneus longus will be measured the "Time to Onset" - expresses the period that passes from the beginning of the fall to the initial recruitment of the Peroneus longus.
Electromyography of peroneus longus- "The height of the amplitude"-unexpected fall | Within 24 hours
  Subjects will stand on a platform during a unilateral sudden 30° inversion platform perturbation that resembles an unexpected fall. electromyography of peroneus longus will be measured the "height of the amplitude" - expresses the peak of the electrical activity of the Peroneus longus muscle.
Electromyography of peroneus longus- "Time to Peak"-unexpected fall | Within 24 hours
  Subjects will stand on a platform during a unilateral sudden 30° inversion platform perturbation that resembles an unexpected fall. electromyography of peroneus longus will be measured the "Time to Peak"- describes the time it takes for the Peroneus longus muscle to reach the peak of its electrical activity.
Electromyography of peroneus longus- "Time to Onset"-unexpected fall | Within 24 hours
  Subjects will stand on a platform during a unilateral sudden 30° inversion platform perturbation that resembles an unexpected fall. electromyography of peroneus longus will be measured the "Time to Onset"- expresses the period that passes from the beginning of the fall to the initial recruitment of the Peroneus longos muscle.
Maximal voluntary isometric peroneal contraction force | Within 24 hours
  Subject will perform Maximal voluntary isometric peroneal contraction. The force will measured with dynamometer

CONTACTS AND LOCATIONS:
Locations (1):
- Ariel University -The Neuromuscular & Human performance laboratory, Ariel, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hayek R, Gottlieb U, Gutman I, Springer S. Peroneal muscle response to single-leg drop-jump and unexpected leg-drop in young and middle-aged adults before and after one session of neuromuscular training. Eur Rev Aging Phys Act. 2023 Jun 17;20(1):11. doi: 10.1186/s11556-023-00321-8. PMID 37330500